CLINICAL TRIAL: NCT05424484
Title: Mesh Augmented Reinforcement of Abdominal Wall Suture Line in Patients Undergoing Midline Laparotomy to Limit the Rate of Incisional Hernia Occurrence
Brief Title: Mesh Augmented Reinforcement of Abdominal Wall Suture Line to Limit the Rate of Incisional Hernia Occurrence
Acronym: MARS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MDT20049MARS; CIV-22-05-039590 (Other: Eudamed)
Record Dates: First submitted 2022-05-18; First posted 2022-06-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Incisional Hernia; Incisional Hernia of Midline of Abdomen; Midline Laparotomy
Keywords: Incisional Hernia; Prophylactic Mesh; Incisional Hernia of Midline of Abdomen; Midline Laparotomy
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hernia prevention cohort (Experimental): single arm study, no control arm
  Interventions: Device: Self-Gripping Resorbable Mesh

INTERVENTIONS:
Device: Self-Gripping Resorbable Mesh — Self-Gripping Resorbable Mesh used for suture line reinforcement after midline laparotomy in clean and clean-contaminated fields (CDC Classification I and II).

SUMMARY:
The purpose of this prospective, pivotal, multi-center, single-arm, pre-market, investigational clinical study is to assess the safety and performance of Deternia™ Self-Gripping Resorbable Mesh when used for suture line reinforcement after midline laparotomy in clean and clean-contaminated fields (CDC Classification I and II). Data from this study will be used to support market applications. The indication under investigation is reinforcement of midline laparotomy to limit the rate of incisional hernia (IH) in clean and clean-contaminated surgeries (CDC Classification I and II).

DETAILED DESCRIPTION:
The primary objective of this investigation is to evaluate the performance of Deternia™ Self-Gripping Resorbable Mesh when used for suture line reinforcement after elective midline laparotomy in clean and clean-contaminated fields (CDC Classification I and II) at 12 months post-operatively and to demonstrate expected performance in terms of rate of IH occurrence relative to a performance goal (based on historical data on primary laparotomy incision suture closure with small bites only).

The secondary objectives are to evaluate the safety and performance of Deternia™ Self-Gripping Resorbable Mesh when used for suture line reinforcement after elective midline laparotomy in clean and clean contaminated fields (CDC Classification I and II) within 36 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent.
2. Subject is ≥18 years of age at the time of consent.
3. Subject will be undergoing an elective surgery with a planned/possible midline laparotomy with retrorectus mesh placement.

3a. Subject will be undergoing an elective laparoscopy with a planned possibility of a conversion to midline laparotomy or an elective laparoscopy with a planned possible midline laparotomy for specimen extraction.

Pre-Operative Exclusion Criteria:

1. Subject is undergoing emergency surgery, i.e. lifesaving procedures performed where patient is in imminent danger of death
2. Subject has a history of allergic reactions after application of poly-L-lactide, poly-trimethylene carbonate copolymers (PLLA/TMC)
3. Subject is pregnant or is planning pregnancy during study duration period (Females of child-bearing potential will be required to provide either a urine or serum pregnancy test (except for subjects who are surgically sterile or are at least 2 years postmenopausal)) 3a. Subject is breastfeeding or is planning to breastfeed during the study duration period
4. Subject is unable or unwilling to comply with the study requirements or follow-up schedule
5. Subject is scheduled for another planned surgery, and subsequent surgery would jeopardize previous application of study treatment
6. Subject with a body mass index (BMI) > 45 kg/m2
7. Subjects with the following medical interventions/medical conditions are excluded from participation in the study: uncontrolled diabetes (hemoglobin A1c (Hb1Ac) > 60mmol/mol), cirrhosis, stoma wearers
8. Concomitant ostomy (stoma creation or closure)
9. Subject who had received a mesh in a previous ventral hernia repair or has an existing ventral hernia > 2 cm
10. Subject with a life expectancy inferior to the study follow-up duration (36 months)
11. Study procedure is a relaparotomy within 30 days of previous abdominal surgery
12. Subject with an American Society of Anesthesiologists (ASA) scores higher than 3
13. Subject has participated in an investigational drug study within the washout period of the drug or in a device study that would interfere with mesh implantation or assessment of Incisional Hernia
14. Subject with current chemo and/or radiation therapy within 2 weeks of procedure

    Only exclusion of chemotherapeutic drugs that have:
    * Cytotoxic effect and/or
    * Inhibit of cell replication and/or
    * Impaired tissue healing
15. Subject with any history of ascites
16. Subject has a medical condition that precludes the patient from participation in the opinion of the investigator
17. Subject is undergoing a vascular procedure other than abdominal aortic aneurysm (AAA) surgery (i.e, only AAA surgeries accepted)

Intraoperative Exclusion criteria

1. Subject's study procedure is in a contaminated or infected site as assessed by the Investigator(s) (CDC Class 3 and 4)
2. Abdomen is left open at the end of the procedure
3. Subject has an unsuspected ventral hernia >2cm encountered at the time of laparotomy
4. Inability to close the anterior fascia or keep the mesh securely out of the peritoneal cavity
5. Second-look procedure planned
6. Cases requiring a full-thickness partial resection of the abdominal wall (in particular the midline) because of involvement in neoplastic process or complex fistula
7. Inoperable tumor/poor prognostic cancer/patient non curatively treated
8. Subject has a suture length to wound length ratio< 3.5/1
9. Subject has any ongoing infection at the time of the surgery, that is uncontrolled and/or requiring treatment such as antibiotics
10. Subject was not implanted with Deternia™ Self Gripping Resorbable Mesh
11. Subject requires more than 1 mesh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incisional Hernia Rate | 12 months
  Occurrence of incisional hernia assessed by clinical examination and abdominal ultrasound exam

SECONDARY OUTCOMES:
Incisional Hernia Rate | 24- and 36-months
  Occurrence of incisional hernia assessed by clinical examination and abdominal ultrasound exam
Incisional Hernia Rate | 3-, 6-, 12-, 24-, and 36- months
  Occurrence of incisional hernia assessed by clinical examination
Time to Incisional Hernia | From the surgery to the 36-month visit
  Time from surgery to incisional hernia
Time to other adverse device effects (ADE) | From the surgery to the 36-month visit
  Time from skin incision to ADE
Incidence of all adverse device effects (ADEs) | Intra-operatively, at discharge (post-surgery up to 3-mo), and within 3-, 6-, 12-, 24-, and 36- months
  Adverse device effects related to mesh and mesh-augmented reinforcement procedure
Incidence of adverse events (AEs) of interest | Intra-operatively, at discharge (post-surgery up to 3-mo), and within 3-, 6-, 12-, 24-, and 36- months
  AEs of interest: symptomatic seroma requiring action taken, hematoma needing surgical revision, surgical site infection (SSI) defined via the CDC classification of SSI (superficial, deep or organ space), wound dehiscence (skin and/or fascial), mesh removal
Pain at the site of surgery evaluated with Numeric Rating Scale (NRS) | baseline (screening), discharge (post-surgery up to 3-mo) and at 3-, 6-, 12-, 24-, and 36- months
  Scale from 0-10, with 0 being no pain and 10 being the worst imaginable pain
EQ-5D-5L quality of life (QoL) | Baseline and at 3-, 6-, 12-, 24-, and 36- months
  Self-administered QOL questionnaire with 5 questions on quality of life and a numeric scale from 0-100 with 0 being the worst health you can imagine and 100 being the best health you can imagine.
Surgeon Satisfaction | Day 0, post-operative
  Surgeon satisfaction questionnaire on mesh use
Hospital length of stay | Hospital admission to hospital discharge (post-surgery up to 3-mo)
  Amount of time spent inpatient
Readmission and reoperation rate | From the surgery to the 36-month visit
  Related to Mesh device and/or Mesh Augmented Reinforcement procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen, MD, Study Chair — Oululu University Hospital, Oululu, Finland
Locations (13):
- Croatia (2):
  - Clinical Hospital Center Sisters of Mercy, Zagreb
  - University Hospital Center of Zagreb, Zagreb
- Germany (3):
  - Klinikum Braunschweig, Braunschweig
  - Pius-Hospital Medical Campus University of Oldenburg, Oldenburg
  - Barmherzige Brüder Regensburg, Regensburg
- Netherlands (2):
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Maastricht University Medical Center, Maastricht
- Spain (4):
  - Consorci Sanitari de l'Anoia Hospital Universitari d'Igualada, Igualada, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (2):
  - Countess Of Chester Hospital NHS Foundation Trust, Chester, Cheshire
  - Cardiff and Vale University Local Health Board, Cardiff

IPD SHARING:
Plan to Share IPD: No